CLINICAL TRIAL: NCT02694185
Title: Secondary Event Prevention Using Population Risk Management After PCI
Brief Title: Secondary Event Prevention Using Population Risk Management After PCI and for Anti-Rheumatic Medications
Acronym: SEPPRMACI-ARM
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Health Services Research
Other Study IDs: IIR 14-048; 16-1419 (Other: CIRB); 1I01HX001604-01A2 (NIH)
Record Dates: First submitted 2016-02-16; First posted 2016-02-29 (Estimated); Results first posted 2021-06-25 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-08

CONDITIONS: Myocardial Ischemia; Rheumatic Diseases
Keywords: Medication Adherence; Randomized Controlled Trial; Veterans
MeSH Terms: conditions — Myocardial Ischemia; Rheumatic Diseases; Medication Adherence

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental Group (Experimental): This group will undergo the intervention as described in the protocol
  Interventions: Other: Caplan IVR
- Control Group (No Intervention): This group will not receive the intervention, they will receive usual care

INTERVENTIONS:
Other: Caplan IVR — This intervention will consist of: proactive real-time adherence monitoring of patients and targeting of individuals only when they have exhibited non-adherence behavior (i.e., if patients have not refilled their medication more than 4 or 7 days after it was due to be refilled). The intervention will employ a tailored, escalating-intensity approach which begins with some combination of personalized short messaging service (SMS) text messages and interactive voice response (IVR) telephone technology, depending on patient preference. Patients failing SMS and then IVR by not refilling their medication (or declining SMS and failing IVR) escalate to a trained research interventionalist (typically, a clinical pharmacist). The interventionalist will contact the patient and address adherence barriers based on the dimensions outlined by the World Health Organization (WHO) that are specific to each patient.
  Arms: Experimental Group

SUMMARY:
Ischemic heart disease (IHD) and its treatment carry profound public health and economic implications. Among Veterans, IHD represents one of the most common causes of death and disability, with over 500,000 affected individuals' annually. Rheumatic disease, though far less common than IHD can affect multiple organ systems and requires therapies costing in excess of $50,000 a year. Optimal treatment of Veterans with IHD and rheumatic disease requires a number of medications to maintain or improve health. Not taking medications as prescribed, however, is common and increases the risk of subsequent adverse events (cardiac death and myocardial infarction [MI]).

To improve medication adherence rates and the cardiac health of Veterans with IHD, the investigators propose to test a medication adherence intervention. Known as VA SEPPRMACI-ARM (Secondary Event Prevention using Population Risk Management After PCI and for Anti-Rheumatic Medications), this intervention will consist of: proactive real-time adherence monitoring of patients and targeting of individuals if they have not refilled their medication a given number of days after it was due for refill. The intervention will employ a tailored, escalating-intensity approach which begins with some combination of personalized short messaging service (SMS) text messages and interactive voice response (IVR) telephone technology, depending on patient preference. Patients not completing SMS and then IVR by not refilling their medication (or declining SMS and not completing IVR) escalate to a trained research interventionalist. The interventionalist will contact the patient and address adherence barriers based on the dimensions outlined by the World Health Organization (WHO) that are specific to each patient. The investigators will test the intervention on IHD patients who have recently undergone PCI-a cardiac procedure commonly used among IHD patients to improve the heart's blood flow and in patients starting anti-rheumatic medication. The investigators will test the intervention at four VA Cardiac Catheterization Laboratories (CCLs) and have 12 sites serving as usual care controls.

DETAILED DESCRIPTION:
Ischemic heart disease (IHD) and rheumatic diseases are both pervasive, expensive, and results in grave health consequences. IHD affects an estimated 15.4 million Americans 20 years of age-representing 6.4% of the adult population. The direct and indirect cost of IHD has been estimated at $195.2 billion, with a doubling of cost projected by 2030.5 Similarly, the direct cost to the U.S. workforce for rheumatoid arthritis alone approaches $5.8 billion yearly.

Widely-accepted national evidence-based guidelines support the use of cardio-protective medications to reduce the risk of adverse consequences resulting from IHD and disease modifying anti-rheumatic medications (DMARDs) to reduce the risk of adverse consequence in rheumatic diseases. For example, numerous rigorously conducted randomized trials show that statins improve outcomes and reduce mortality in patients with established cardiovascular disease (i.e., secondary prevention), including those undergoing percutaneous coronary interventions (PCI). The use of statins and beta-blockers have been repeatedly demonstrated to be cost-effective in lowering cardiovascular event (CVE) rates, in part by their effects on cholesterol, and blood pressure, respectively. Accordingly, the most recent VA performance measures and American Heart Association guidelines encourage the use of statins in patients with atherosclerotic disease; beta-blockers in subjects with left ventricular systolic dysfunction (ejection fraction less than 40%), prior MI, or blood pressure of 140/90 or greater; and clopidogrel following any acute coronary syndrome (ACS) or PCI with stent. The rheumatology literature provides similar evidence for the benefit of DMARDs in rheumatic diseases, and guidelines strongly endorse their use.

Unfortunately, non-adherence to medications is common, and increases the risk of poor outcomes. The investigators' 2011 national preliminary data from VA cardiac catheterization laboratories (CCLs) demonstrate that over 6300 patients experienced at least one refill gap of >= 7 days for statins in the year following PCI. The mean proportion of days covered (PDC) for these patients was only 75%-below the PDC threshold of 80% that typical defines adherent patients, based on the empiric evidence for effectiveness of medications at this cut-point. Non-adherent patients were present at all CCLs without substantial variation in mean PDC by center, suggesting a global problem.

Systematic problems underlie and contribute to non-adherence to medications. Usual care of IHD and rheumatic disease patients is encumbered by systematic deficiencies including: passive monitoring (contact with patients only when initiated by the patient) and inefficiency (time-consuming patient-by-patient approach, rather than through population management). The proposed intervention addresses both the complex patient-specific factors (emphasizing forgetfulness and carelessness) and the systematic inadequacies using a multi-modal, escalating approach.

Objectives

1. To assess the effectiveness of a multi-faceted patient-centered intervention versus usual care in improving medication adherence as measured by proportion of days covered (PDC, primary outcome). This will be tested among IHD patients for statins, beta-blockers and clopidogrel in the year after PCI and among rheumatology clinic patients chronically prescribed DMARDs. Hypothesis: The PDC for patients in the intervention arm will exceed the PDC for the usual care arm by a 10% absolute difference.
2. (Secondary outcome): To determine the effectiveness of a multi-faceted patient-centered intervention versus usual care in reducing secondary CVEs (myocardial infarction [MI], repeat revascularization [PCI or coronary bypass graft], and all-cause mortality) among IHD patients at 18 months post-PCI and progressive erosive disease demonstrated on plain film radiographs in patients with rheumatic diseases (i.e. "radiographic progression"). Hypothesis: The rate of CVEs and radiographic progression will be 5% relatively lower for patients in the intervention arm compared with usual care.
3. (Secondary outcome): To establish the cost to implement and maintain the intervention, above the cost of usual care, as well as the incremental cost effectiveness (ICE; e.g. cost to achieve at 10% improvement in PDC; cost per CVE prevented). Hypothesis: This aim does not posit a hypothesis as the objective is descriptive. The available funding for this project limits this outcome to IHD patients (no rheumatic disease patients will be analyzed according to cost).

ELIGIBILITY:
Inclusion Criteria:

Patients will qualify for inclusion if they:

1. Undergo PCI or are prescribed a DMARD.
2. Are prescribed any of the following medications:

   [for the IHD intervention]
   * Statin
   * Beta-blocker
   * Thienopyridines (dual platelet inhibitors)

   [for the DMARD intervention]
   * Oral methotrexate
   * Sulfasalazine
   * Azathioprine
   * Leflunomide
   * Tofacitinib
   * Hydroxychloroquine [Note: as a study focused on adherence, the investigators will NOT address the appropriateness of prescribed medications, which is an important, but separate issue]
3. Receive their care from the VA. This is defined by the presence of a VA-assigned-PCP in the year prior to PCI or in the year following PCI (IHD intervention) or in the year prior to or following index DMARD prescription (rheumatic disease intervention).

Exclusion Criteria:

Patients will be excluded under the following circumstances:

* Undergoing only diagnostic (non-interventional) catheterization
* Receive their index medicines (listed in item above) from a non-VA source
* Discharge to nursing home or skilled nursing facility
* Individuals with impaired decision making capacity
* Prisoners
* Pregnant women
* The terminally ill

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5269 (Actual)
Dates: Start 2016-10-01 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2025-02-28 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Liron Caplan, MD PhD, Principal Investigator — Rocky Mountain Regional VA Medical Center, Aurora, CO
Locations (5):
- United States (4):
  - San Francisco VA Medical Center, San Francisco, CA, San Francisco, California
  - Rocky Mountain Regional VA Medical Center, Aurora, CO, Aurora, Colorado
  - Baltimore VA Medical Center VA Maryland Health Care System, Baltimore, MD, Baltimore, Maryland
  - Durham VA Medical Center, Durham, NC, Durham, North Carolina
- VA Caribbean Healthcare System, San Juan, PR, San Juan, Puerto Rico

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Raghavan S, Liu WG, Michael Ho P, Plomondon ME, Baron AE, Caplan L, Joynt Maddox KE, Magid D, Saxon DR, Voils CI, Bradley SM, Maddox TM. Coronary artery disease severity modifies associations between glycemic control and both mortality and myocardial infarction. J Diabetes Complications. 2018 May;32(5):480-487. doi: 10.1016/j.jdiacomp.2018.01.010. Epub 2018 Jan 31. PMID 29483016
- [Background] Baker JF, Sauer B, Teng CC, George M, Cannon GW, Ibrahim S, Cannella A, England BR, Michaud K, Caplan L, Davis LA, O'Dell J, Mikuls TR. Initiation of Disease-Modifying Therapies in Rheumatoid Arthritis Is Associated With Changes in Blood Pressure. J Clin Rheumatol. 2018 Jun;24(4):203-209. doi: 10.1097/RHU.0000000000000736. PMID 29664818
- [Background] Yazdany J, Caplan L, Fitzgerald J, Schmajuk G. Editorial: The Evolving Art and Science of American College of Rheumatology Guidelines. Arthritis Rheumatol. 2019 Jan;71(1):2-4. doi: 10.1002/art.40725. Epub 2018 Nov 30. No abstract available. PMID 30499229
- [Background] McCulley CB, Barton JL, Cannon GW, Sauer BC, Teng CC, George MD, Caplan L, England BR, Mikuls TR, Baker JF. Body mass index and persistence of conventional DMARDs and TNF inhibitors in rheumatoid arthritis. Clin Exp Rheumatol. 2019 May-Jun;37(3):422-428. Epub 2018 Nov 7. PMID 30418120
- [Background] Hirsh J, Wood P, Keniston A, Boyle D, Quinzanos I, Caplan L, Davis L. Universal Health Literacy Precautions Are Associated With a Significant Increase in Medication Adherence in Vulnerable Rheumatology Patients. ACR Open Rheumatol. 2020 Feb;2(2):110-118. doi: 10.1002/acr2.11108. Epub 2020 Jan 19. PMID 31957348
- [Background] Raghavan S, Liu WG, Berkowitz SA, Baron AE, Plomondon ME, Maddox TM, Reusch JEB, Ho PM, Caplan L. Association of Glycemic Control Trajectory with Short-Term Mortality in Diabetes Patients with High Cardiovascular Risk: a Joint Latent Class Modeling Study. J Gen Intern Med. 2020 Aug;35(8):2266-2273. doi: 10.1007/s11606-020-05848-5. Epub 2020 Apr 24. PMID 32333313
- [Background] Daniel CM, Davila L, Makris UE, Mayo H, Caplan L, Davis L, Solow EB. Ethnic Disparities in Atherosclerotic Cardiovascular Disease Incidence and Prevalence Among Rheumatoid Arthritis Patients in the United States: a Systematic Review. ACR Open Rheumatol. 2020 Sep;2(9):525-532. doi: 10.1002/acr2.11170. Epub 2020 Sep 1. PMID 32869533

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study will employ an approach to consent similar to SDP-179 Hybrid Effectiveness-Implementation Study to Improve Clopidogrel Adherence which has previously been approved by (CIRB Protocol #12-12). The study will enroll all subjects undergoing PCI or using DMARDs at 16 VA Medical Centers. These Medical Centers are all tertiary referral hospitals within their respective VISN and provide a full spectrum of cardiac and rheumatologic care services.
Period: Overall Study
Arm/Group | Experimental Group | Control Group
Started | 476 | 4793
Completed | 431 | 4793
Not Completed | 45 | 0
Not completed — Withdrawal by Subject | 45 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Experimental Group | Control Group | Total
Number analyzed (Participants) | 431 | 4793 | 5224
Age, Continuous [Mean (Full Range); unit: years] | 68.6 [62.9 to 73.1] | 68.7 [63.0 to 72.6] | 68.7 [62.9 to 73.1]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 103 | 115
  Male | 419 | 4690 | 5109
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 330 | 3789 | 4119
  African American | 89 | 872 | 961
  Other | 12 | 132 | 144
Region of Enrollment [Count of Participants; unit: Participants]
  Puerto Rico | 42 | 214 | 256
  United States | 389 | 4579 | 4968

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Days Covered (PDC)
Description: Proportion of Days Covered (PDC) is measured by looking at the number of doses of medication a patient has versus days in the month (if a patient has 20 days of medication for a 30 day period their PDC is 20/30, 2/3, or 66.7%). Used to assess the effectiveness of the intervention, PDC will be tested among IHD patients in the year after PCI and among rheumatology clinic patients chronically prescribed DMARDs.
Time Frame: 1 year
Population: Participant numbers differ below because not all subjects are taking an anti-platelet, beta-blocker, and statin medication.
Measure: Mean (95% Confidence Interval); unit: percentage of days covered
Arm/Group | Experimental Group | Control Group
Number analyzed (Participants) | 431 | 4793
percentage of days covered
  Anti-platelet: number analyzed (Participants) | 421 | 4691
  Anti-platelet | 82.6 [77.9 to 86.2] | 75.6 [69.7 to 79.9]
  Beta-Blocker: number analyzed (Participants) | 315 | 3924
  Beta-Blocker | 78.4 [71.5 to 82.7] | 73.3 [66.8 to 77.1]
  Statin: number analyzed (Participants) | 327 | 4250
  Statin | 78.8 [71.8 to 83.4] | 71.2 [64.9 to 75.1]

2. Secondary Outcome: Cardiovascular Events (CVE)
Description: Cardiovascular Events (CVEs) such as mortality, myocardial infarction, stroke, or repeat revascularization among IHD patients at 12 months post-PCI and progressive erosive disease demonstrated in patients with rheumatic disease will be monitored. CVEs will be monitored to determine if there is a reduction in the occurrence of those events as a result of the intervention.
Time Frame: 1 year
Measure: Mean (95% Confidence Interval); unit: Cardiovascular events
Arm/Group | Experimental Group | Control Group
Number analyzed (Participants) | 431 | 4793
Cardiovascular events | 15.2 [10.9 to 25.5] | 14.3 [12.3 to 16.7]

3. Secondary Outcome: Incremental Cost Effectiveness (ICE)
Description: To establish the cost to implement and maintain the intervention, above the cost of usual care. Incremental Cost Effectiveness (ICE) is the cost to achieve a 10% improvement in PDC, and the cost of CVE prevented.
Time Frame: through study completion, an average of 1 year
Measure: Median (Inter-Quartile Range); unit: dollars per patient
Arm/Group | Experimental Group | Control Group
Number analyzed (Participants) | 431 | 4793
dollars per patient | 821.45 [158.18 to 1541.91] | 893.55 [437.85 to 1460.85]

ADVERSE EVENTS:
Time Frame: Adverse event data were collected beginning from enrollment to study completion; average duration per participant was one year, per the design of the study.
Description: Over the duration of the entire study, there have been 23 patients who passed away in the intervention group. The Data Safety Monitoring Board did not attribute any deaths to their participation in the research or the intervention.
Arm/Group | Experimental Group | Control Group
All-Cause Mortality (participants affected / at risk) | 23/476 | 209/4793
Serious Adverse Events (participants affected / at risk) | 0/476 | 0/4793
Other Adverse Events (participants affected / at risk) | 0/476 | 0/4793

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-03-06): https://cdn.clinicaltrials.gov/large-docs/85/NCT02694185/Prot_SAP_000.pdf